CLINICAL TRIAL: NCT05303662
Title: Prevalence of Multidrug Resistant Micro-organism Carriage in Patients Undergoing an Endoscopic Retrograde Cholangiopancreatography in Four Different Countries
Brief Title: Prevalence of Multidrug Resistant Micro-organism Carriage in Patients Undergoing an ERCP in Four Different Countries
Acronym: PREVENT
Status: Completed | Type: Observational
Sponsor: Marco J. Bruno (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Marco J. Bruno, Professor of Gastroenterology and Hepatology, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: NL79136.078
Record Dates: First submitted 2022-03-17; First posted 2022-03-31 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Drug Resistance, Multiple, Bacterial; Cholangiopancreatography, Endoscopic Retrograde
Keywords: Cholangiopancreatography, Endoscopic Retrograde; Drug Resistance, Multiple, Bacterial; Equipment Contamination; Duodenoscope associated infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Only in the Netherlands biospecimen retention will take place to study secondary objectives: feces, urine, wound tissue, blood, bile, rectal swabs, duodenal aspirate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- ERCP-patients Netherlands: Patients undergoing ERCP in the study site in the Netherlands
  Interventions: Diagnostic Test: Multidrug-Resistant Organisms (MDRO) testing through rectal and oral/nasal swabs; Diagnostic Test: MDRO-testing duodenal aspirate; Diagnostic Test: Microbiome through rectal swab; Diagnostic Test: Microbiome testing duodenal aspirate
- ERCP-patients Italy: Patients undergoing ERCP in the study site in Italy
  Interventions: Diagnostic Test: Multidrug-Resistant Organisms (MDRO) testing through rectal and oral/nasal swabs
- ERCP-patients United States: Patients undergoing ERCP in the study site in the Netherlands
  Interventions: Diagnostic Test: Multidrug-Resistant Organisms (MDRO) testing through rectal and oral/nasal swabs
- ERCP-patients India: Patients undergoing ERCP in the study site in India
  Interventions: Diagnostic Test: Multidrug-Resistant Organisms (MDRO) testing through rectal and oral/nasal swabs; Diagnostic Test: MDRO-testing duodenal aspirate

INTERVENTIONS:
Diagnostic Test: Multidrug-Resistant Organisms (MDRO) testing through rectal and oral/nasal swabs — Pooled throat/nose sample and a rectal sample is taken prior to the ERCP
Diagnostic Test: MDRO-testing duodenal aspirate — Duodenal aspirate is collected from the duodenum, diluted and undiluted. Then cultured for presence of MDRO's
  Groups: ERCP-patients India; ERCP-patients Netherlands
Diagnostic Test: Microbiome through rectal swab — An rectal swab is collected for microbiome purposes
  Groups: ERCP-patients Netherlands
Diagnostic Test: Microbiome testing duodenal aspirate — Duodenal aspirate is collected from the duodenum, diluted and undiluted for microbiome analysis
  Groups: ERCP-patients Netherlands

SUMMARY:
The duodenoscopes currently used for Endoscopic Retrograde Cholangio - and Pancreaticography (ERCP) examinations are reusable and are therefore washed and disinfected after each use. Despite this, these endoscopes sometimes remain contaminated with bacteria. Several reports of outbreaks linked to contaminated duodenoscopes have been published worldwide. Recently, the Food and Drug Administration (FDA) advised manufacturers and health care professionals to transition away from fixed endcap duodenoscopes and instead focus more on the use of duodenoscopes with disposable components or fully disposable duodenoscopes. Single-use endoscopes have been developed, but they are not yet widely used, partly because of the extra costs that these endoscopes add to the examination. A possible interim solution, is to only use these disposable endoscopes in patients who carry multi-resistant bacteria in order to prevent the spread of these bacteria. For this, it is important to know how many people who undergo an ERCP carry multi-resistant bacteria. The primary objective of this study is to measure the prevalence of multi-resistant bacteria in patients undergoing ERCP in four different countries: India, the Netherlands, Italy and the United States. In the Netherlands, some secondary outcomes will be investigated with regard to the prevalence of duodenoscope contamination, the risk of bacterial transmission via a contaminated duodenoscope and the presence of multi-resistant bacteria in the duodenum.

ELIGIBILITY:
Inclusion Criteria:

* The subject is planned to undergo an ERCP procedure, either through an outpatient department or an inpatient department
* The subject is capable to understand the information required to give informed consent

Exclusion Criteria:

* In case the inclusion criteria were not met

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ERCP procedures irrespective of the indication for that procedure
Sampling Method: Probability Sample
Enrollment: 1244 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of multidrug resistant micro-organism carriage in patients undergoing an ERCP in four different countries | 1 week
  Prevalence (as a percentage) of Methicillin-resistant Staphylococcus aureus (MRSA) in nasal or throat swabs, along with rectal carriage rates of Extended Spectrum Beta-Lactamase (ESBL), Vancomycin-resistant Enterococci (VRE), Carbapenem-resistant Enterobacterales (CRE), Carbapenemase-Producing Pseudomonas aeruginosa (CPP), and resistant Acinetobacter among ERCP patients in India, the Netherlands, Italy, and the United States.

SECONDARY OUTCOMES:
Prevalence of multidrug resistant micro-organism carriage in the duodenum of patients undergoing ERCP compared to the rectum | 1 week
  Prevalence (as a percentage) of duodenal carriage of MRSA, ESBL, VRE, CRE, CPP, and resistant Acinetobacter among ERCP patients in both India and the Netherlands.
Differences of rectal microbiome between ERCP patients carrying MDRO compared to patients without MDRO | 1 week
  Sequencing data analysis, such as 16S rRNA gene sequencing, will be used to assess the overall composition of the rectal microbiome. This will involve the identification of various bacterial taxa present in the samples and determining their relative proportions. The results will provide information on the broader microbial community composition.
  These results will be compared between ERCP patients carrying MDRO and those without MDRO to investigate differences in both specific bacterial species' abundance and overall microbiome composition.
Prevalence of duodenoscope-associated infections and colonizations | 6 months
  Comparison of isolates form duodenoscope cultures with isolates from clinical cultures from patients treated with a contaminated duodenoscope in order to detect transmission.
Differences of duodenal microbiome between ERCP patients carrying MDRO compared to patients without MDRO | 1 week
  Sequencing data analysis, such as 16S rRNA gene sequencing, will be used to assess the overall composition of the duodenal microbiome. This will involve the identification of various bacterial taxa present in the samples and determining their relative proportions. The results will provide information on the broader microbial community composition.
  These results will be compared between ERCP patients carrying MDRO and those without MDRO to investigate differences in both specific bacterial species' abundance and overall microbiome composition.

CONTACTS AND LOCATIONS:
Overall Officials: M. J. Bruno, Professor, Principal Investigator — Erasmus Medical Center
Locations (4):
- UPMC, Pittsburgh, Pennsylvania, United States
- AIG hospitals, Hyderabad, Telangana, India
- Humanitas research hospital, Milan, Lombardy, Italy
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rauwers AW, Voor In 't Holt AF, Buijs JG, de Groot W, Hansen BE, Bruno MJ, Vos MC. High prevalence rate of digestive tract bacteria in duodenoscopes: a nationwide study. Gut. 2018 Sep;67(9):1637-1645. doi: 10.1136/gutjnl-2017-315082. Epub 2018 Apr 10. PMID 29636382
- [Derived] van der Ploeg K, Vos MC, Rughwani H, Severin JA, Post RAJ, Reddy DN, Veturi SY, Sasikala M, Memon SF, Repici A, Spadaccini M, Colombo M, Andreozzi M, Stevens BA, Das R, Slivka A, Mason-Slingerland BCGC, Bruno MJ. Preprocedural screening for multidrug-resistant organisms in endoscopic retrograde cholangiopancreatography: an international, multicentre, cross-sectional observational study. EClinicalMedicine. 2025 Nov 13;90:103627. doi: 10.1016/j.eclinm.2025.103627. eCollection 2025 Dec. PMID 41324017